CLINICAL TRIAL: NCT03439150
Title: Recovery of Microvascular Myocardial Resistance After ST Elevation Myocardial Infarction and Its Relation to Outcome. A Prospective Exploratory Study
Brief Title: Resistance STEMI Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrolment
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Nico Pijls, N.H.J Pijls, MD, PhD, Professor of Cardiology, Catharina Ziekenhuis Eindhoven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Resistance STEMI
Record Dates: First submitted 2018-02-02; First posted 2018-02-20 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: STEMI; Acute Myocardial Infarction
Keywords: Absolute flow measurement; Microvascular resistance; Left ventricular function
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study arm (Other): The study arm will undergo absolute flow and resistance measurements immediately after PPCI of the culprit artery
  Interventions: Diagnostic Test: Absolute flow and resistance measurement

INTERVENTIONS:
Diagnostic Test: Absolute flow and resistance measurement — Absolute flow and resistance measurements immediately after PPCI of the culprit vessel (in a STEMI setting) and repeated absolute flow and resistance measurements after 3-7 days

SUMMARY:
In acute myocardial infarction, early restoration of blood flow to the jeopardized myocardium is of paramount importance to limit infarct size and to improve long term outcome. Primary percutaneous coronary intervention (PPCI) is the treatment of choice in these patients. Despite achievement of adequate epicardial coronary artery reperfusion in many patients, transient or persistent myocardial microvascular dysfunction is often present, also referred to as the no-reflow phenomenon. This microvascular dysfunction and the time course during which it recovers, is most likely also related to long term outcome.

If microvascular reperfusion is still limited immediately after myocardial infarction but recovers quickly in the days thereafter, this might be beneficial for long term prognosis.

Several treatments have been suggested to limit microvascular injury and to improve microvascular reperfusion in the acute phase of myocardial infarction (such as intra-aortic balloon pumping, glycoprotein IIB/IIIA inhibitors, adenosine, verapamil, nitroglycerine, cyclosporine, or gap-junction-inhibitors), but it has been difficult to assess the effect of such treatment due to the simple fact that no methodology has been available for quantitative assessment of the microcirculation of the heart.

Assessment of microvascular perfusion and function has been very difficult so far and has been hampered by a number of methodological and technical shortcomings. Measurement of absolute blood flow in the infarcted area and true quantitative calculation of absolute resistance in acute myocardial infarction, has been introduced in the last years using a technique with thermodilution and continuous infusion of small amounts of saline. This technique offers the possibility to study the course of microvascular (dys)function after acute myocardial infarction with potentially important implications for treatment at follow-up. Technical performance of such measurements was difficult so far because of a complex instrumentation and the necessity of additional administration of intravenous adenosine. In the last 2 years, this technique has been largely simplified by the introduction of a new multipurpose monorail infusion catheter (RayFlow ®, Hexacath, Paris) and the observation that saline infusion of 15-20 ml/min in itself already ensures maximum coronary hyperemia. Finally, easy to handle software has been developed for online interpretation of such measurements. Consequently, measurement of absolute blood flow and myocardial resistance has become easy to perform now and the complete measurements only take a few minutes in addition to a regular PPCI or Fractional Flow Reserve (FFR) measurement. The measurements are absolutely safe, reproducible, only a small amount of saline (100 ml at room temperature) is needed, no additional medication is necessary, the patient doesn't experience any discomfort of the measurement and the measurements can be repeated multiple times within minutes.

Therefore, a window is opened for further examination and quantitative assessment of the microcirculation of the heart. The purpose of the present study is to evaluate changes in myocardial resistance over time in ST-Elevation Myocardial Infarction (STEMI) patients, both in the early stage and the subacute phase. Furthermore, the course of such changes and recovery of the microcirculation will be correlated to long-term outcome as assessed by Magnetic Resonance Imaging (MRI) measurements and final infarct size. It is hypothesized that patients can be divided into 3 groups:

A. Patients with an (almost) normal resistance and flow immediately after PPCI B. Patients with still elevated resistance and decreased flow immediately after PPCI, but (partial) recovery in the next days C. Patients with elevated resistance and decreased flow immediately after PPCI which do not recover at all.

The investigators would like to evaluate changes in microvascular resistance of the infarcted area in the first hour after ST-elevation myocardial infarction and during the recovery period (<5 days). Classify patients according to recovery of microvascular resistance and relate the (recovery of) microvascular resistance to outcome and preservation of left ventricular function (with MRI, echo and clinical follow-up at 1 year).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Presentation within 12 hours after the onset of complaints
* Acute ST-elevation myocardial infarction with a total ST segment deviation ≥5 mm
* Able to give and understand informed consent
* Culprit lesion in a proximal or mid-segment of one of the major coronary arteries (diameter ≥2,5 mm), which is stented successfully
* Stable condition after stenting
* One or more additional lesions in one or more different coronary arteries, mandating FFR measurement +/- PPCI during the subacute phase

Exclusion Criteria:

* Age < 18 years or > 75 years
* Cardiogenic shock or pre-shock, determined by the clinician
* Patients with previous myocardial infarction in the culprit artery or with previous bypass surgery
* Very tortuous or calcified coronary arteries
* Long or complex PPCI
* Severe concomitant disease or conditions with a life expectancy of less than 1 year
* Inability to understand and give informed consent
* Known myocardial diseases such as severe left ventricular hypertrophy or cardiomyopathy
* Pregnancy
* Severe conduction disturbances necessitating implantation of a temporary pacemaker
* Contraindications for MRI (claustrophobia, ferromagnetic metal fragments in the body)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Primary endpoint - changes in microvascular resistance | From date of randomization until the date of the second measurements (all within the first week after the index event).
  To evaluate changes in microvascular resistance of the infarcted area in the first hour after ST-elevation myocardial infarction and during the recovery period (<5 days) measured invasively with the absolute flow and resistance measurement.
Co-primary endpoint - risk stratification | From date of randomization until the date of clinical follow-up at 1 year.
  The co-primary endpoint is to see whether the microvascular resistance can classify the patients into groups and identify those with a higher risk of reduced left ventricular function and more adverse events in the end.

SECONDARY OUTCOMES:
Secondary endpoint - left ventricular function | From date of randomization until the date of clinical follow-up at 1 year.
  To relate (recovery of) microvascular resistance to the preservation of left ventricular function (assessed by MRI and echocardiography).
Secondary outcome- Major adverse events | From date of randomization until the date of clinical follow-up at 1 year.
  To relate (recovery of) microvascular resistance to the outcome (adverse events / mortality) during to complete clinical follow up of the patient at 3 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nico Pijls, MD, PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided